CLINICAL TRIAL: NCT00195286
Title: Study of the Safety and Efficacy of Piperacillin/Tazobactam in the Treatment of Patients With Complicated Urinary Infections.
Brief Title: Study Evaluating Piperacillin/Tazobactam in Complicated Urinary Infections.
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 101315
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Urinary Infections
Keywords: Urinary Infections
MeSH Terms: interventions — Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: piperacillin/tazobactam

SUMMARY:
The primary objective is to study the efficacy of piperacillin/tazobactam in patients with complicated urinary tract infections

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients over 16 years of age with complicated urinary infection produced by bacteria that are suspected to be susceptible to treatment with Piperacillin-tazobactam.

Exclusion Criteria:

* Patients known, or thought to be hypersensitivity to beta-lactams
* Patients with an uncomplicated urinary tract infection

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated at internal medicine units
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2004-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (27):
- Spain (27):
  - Antequera (Málaga)
  - Ávila
  - Barcelona
  - Berga (Barcelona)
  - Cadiz
  - Castellon
  - Cáceres
  - Ciudad Real
  - Cuenca
  - Ferrol
  - Granada
  - Jaén
  - Las Palmas
  - Lleida
  - Lorca (Murcia)
  - Lugo
  - Madrid
  - Osuna (Sevilla)
  - Palma Mallorca
  - Pamplona
  - Pontevedra
  - Terrassa
  - Torrelavega
  - Valencia
  - Valladolid
  - Vitoria-Gasteiz
  - Zaragoza